CLINICAL TRIAL: NCT00814593
Title: Randomized Phase II Trial of Intralesional Lymphokine Activated Killer Cells or Polifeprosan 20 With Carmustine Implant (Gliadel® Wafer) as Consolidation Therapy After Primary Treatment of Newly Diagnosed Resectable Glioblastoma
Brief Title: Lymphokine-Activated Killer Cells or Gliadel Wafer in Treating Patients With Newly Diagnosed Glioblastoma Multiforme That Can Be Removed by Surgery
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Hoag Hospital ceased support.
Sponsor: Lisata Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000630437; HOAG-HCC-08-01 (Other: Hoag Cancer Center at Hoag Memorial Hospital Presbyterian)
Record Dates: First submitted 2008-12-24; First posted 2008-12-25 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult giant cell glioblastoma; adult gliosarcoma; adult glioblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Carmustine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Patients undergo intracranial placement of polifeprosan 20 with carmustine implant (Gliadel® wafer) at the time of therapeutic craniotomy.
  Interventions: Drug: polifeprosan 20 with carmustine implant
- Arm II (Experimental): Patients undergo leukapheresis to obtain autologous lymphokine-activated killer (LAK) cells, followed 3-7 days later by therapeutic craniotomy. The autologous LAK cells are then instilled into the tumor bed cavity at the time of therapeutic craniotomy.
  Interventions: Biological: lymphokine-activated killer cells

INTERVENTIONS:
Biological: lymphokine-activated killer cells — Instilled into the tumor bed cavity
  Arms: Arm II
Drug: polifeprosan 20 with carmustine implant — Intracranial placement
  Arms: Arm I

SUMMARY:
RATIONALE: Biological therapies, such as lymphokine-activated killer cells, may stimulate the immune system in different ways and stop tumor cells from growing. Drugs used in chemotherapy, such as Gliadel wafer, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known whether lymphokine-activated killer cells are more effective than Gliadel wafer in treating patients with glioblastoma multiforme.

PURPOSE: This randomized phase II trial is studying the side effects and how well lymphokine-activated killer cells work compared with Gliadel wafer in treating patients with newly diagnosed glioblastoma multiforme that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* To compare the side effects, including infections and/or abnormal healing at the surgery site, associated with intralesional lymphokine-activated killer (LAK) cells vs polifeprosan 20 with carmustine implant (Gliadel® wafer) as consolidation therapy for patients with newly diagnosed resectable glioblastoma multiforme.
* To compare the overall survival of patients treated with these regimens.

OUTLINE: Patients are stratified according to age (< 50 vs ≥ 50 years of age), Karnofsky performance status (70-80% vs 90-100%), use of corticosteroids > 4 mg/day (yes vs no), and progressive disease during first-line therapy (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo intracranial placement of polifeprosan 20 with carmustine implant (Gliadel® wafer) at the time of therapeutic craniotomy.
* Arm II: Patients undergo leukapheresis to obtain autologous lymphokine-activated killer (LAK) cells, followed 3-7 days later by therapeutic craniotomy. The autologous LAK cells are then instilled into the tumor bed cavity at the time of therapeutic craniotomy.

After completion of study treatment, patients are followed periodically for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary malignant glioblastoma multiforme (GBM) (i.e., grade IV anaplastic astrocytoma)
* Must have undergone standard primary therapy (e.g., surgery, radiotherapy, and temozolomide) within the past 90 days

  * Additional anticancer therapy as part of first-line therapy, including a radiosurgical procedure (e.g., stereotactic or gamma knife radiosurgery) allowed
* Must be an operable candidate and willing to undergo craniotomy

PATIENT CHARACTERISTICS:

* Karnofsky performance status 70-100%
* Life expectancy ≥ 2 months
* Hemoglobin > 10.0 g/dL
* AGC > 1,500/mm³
* Platelet count > 100,000/mm³
* Serum total bilirubin < 1.5 times upper limit of normal (ULN)
* ALT and AST < 2.5 times ULN
* Serum creatinine < 1.5 times ULN
* Negative pregnancy test
* Resides in the United States of America
* Venous access available for leukapheresis procedure to obtain peripheral blood mononuclear cells
* No diagnosis of any other invasive cancer within the past 5 years, except in situ carcinoma or basal cell carcinoma or localized squamous cell carcinoma of the skin

  * Patients with prior diagnosis of minimal microscopic cancer (e.g., colonic polyp or stage I prostate cancer with Gleason score < 6) may be eligible, as determined by the principal investigator
* No concurrent serious medical or psychiatric illness that may interfere with giving informed consent or conducting this study
* No known hypersensitivity or allergy to either carmustine or aldesleukin

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 3 weeks since prior anticancer therapy and recovered
* No polifeprosan 20 with carmustine implant (Gliadel® wafer) at the time of prior surgery for GBM
* No prior treatment for progressive disease
* No other concurrent anticancer therapy (e.g., continuation of hormonal therapy for breast or prostate cancer that was diagnosed > 5 years ago)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-11; Primary Completion 2011-04 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Overall survival | 5 years or death, whichever came first.

SECONDARY OUTCOMES:
Rate of significant surgical wound infection (grade 3 or 4) | 4 weeks from date of study treatment.
Rate of grade 3 or 4 non-infectious wound complications | 4 weeks from date of study treatment.
Toxicity as assessed by NCI CTCAE version 3.0 | 4 weeks from date of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Robert O. Dillman, MD, FACP, Principal Investigator — Caladrius Biosciences
Locations (1):
- Hoag Cancer Institute at Hoag Memorial Hospital Presbyterian, Newport Beach, California, United States